CLINICAL TRIAL: NCT01238900
Title: Prospective Evaluation of the Clinical Utility of Placement of Metal Stent for Benign Biliary Strictures
Brief Title: Evaluation of the Use of Metal Stents as Part of the Treatment of Benign Biliary Strictures
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: Benign Biliary Strictures
Record Dates: First submitted 2010-11-05; First posted 2010-11-11 (Estimated); Results first posted 2015-10-02 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-08

CONDITIONS: Benign Biliary Strictures
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- benign biliary strictures: All patients who have a medical indication for an ERCP to place a stent in their benign biliary strictures
  Interventions: Procedure: Endoscopic Retrograde Cholangiopancreatography (ERCP)

INTERVENTIONS:
Procedure: Endoscopic Retrograde Cholangiopancreatography (ERCP) — Endoscopic Retrograde Cholangiopancreatography (ERCP) with placement of metal stent in the bile duct

SUMMARY:
The purpose of this study is to study the evaluation of the use of metal stents as part of the treatment of benign biliary strictures.

DETAILED DESCRIPTION:
In patients with benign biliary strictures, the use of fully covered self-expandable metal stents (SEMS) has been proposed as an alternative to plastic stenting, but high quality prospective data is sparse. This study was performed to evaluate the long -term effectiveness and safety of a new fully covered SEMS for benign biliary strictures.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years or older
2. Subject has benign biliary stricture
3. Subject must be able to give informed consent

Exclusion Criteria:

1. Any contraindication to Endoscopic Retrograde Cholangiopancreatography (ERCP)
2. The subject is unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have a medical indication for endoscopic therapy of benign biliary stictures and are referred for the procedure as part of their standard medical care will be considered for the study.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2009-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Draganov, MD, Principal Investigator — University of Florida
Locations (1):
- Shands at UF endoscopy center, Gainesville, Florida, United States

REFERENCES:
- [Derived] Wagh MS, Chavalitdhamrong D, Moezardalan K, Chauhan SS, Gupte AR, Nosler MJ, Forsmark CE, Draganov PV. Effectiveness and safety of endoscopic treatment of benign biliary strictures using a new fully covered self expandable metal stent. Diagn Ther Endosc. 2013;2013:183513. doi: 10.1155/2013/183513. Epub 2013 May 11. PMID 23956613

RESULTS

PARTICIPANT FLOW:
Groups:
- Benign Biliary Strictures: Participants underwent Endoscopic Retrograde Cholangiopancreatography (ERCP) with placement of self-expandable metal stents (SEMS) in the bile duct.
Period: 6 Months Post Stent Placement
Arm/Group | Benign Biliary Strictures
Started | 23
Completed | 23
Not Completed | 0
Period: <12 Months Post Stent Removal
Arm/Group | Benign Biliary Strictures
Started | 23
Completed | 18
Not Completed | 5
Not completed — Lost to Follow-up | 4
Not completed — persistent stricture after stenting | 1

BASELINE CHARACTERISTICS:
Arm/Group | Benign Biliary Strictures
Number analyzed (Participants) | 23
Age, Customized [Mean (Full Range); unit: years] | 60 [51 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 23
Stricture etiology [Number; unit: participants]
  Chronic pancreatitis (CP) | 14
  Orthotopic liver transplantation (OLT) | 4
  Idiopathic | 4
  Gallstone related | 1
number of participants with history of prior stenting [Number; unit: participants]
  number with prior stenting | 13
  number with no history of stenting | 10

OUTCOME MEASURES:

1. Primary Outcome: Short Term Success Rate in the Resolution of Biliary Strictures
Description: Short-term success was defined as resolution of the stricture as documented by rapid drainage of contrast out of the proximal biliary tree and easy passage of stone extraction balloon inflated to the size of the proximal bile duct. If the biliary stricture had resolved at the 6-month follow-up ERCP, patients were classified as short-term success. If stricture was not resolved at 6-month ERCP then a new SEMS was placed; if the stricture had resolved at the time of the second stent removal, the patient was also classified as short-term success.
Time Frame: 6 months
Population: Of the 23 participants that entered the study, 22 saw short-term success. The population consisted of 14 Chronic pancreatitis patients, 4 postorthotopic liver transplant patients, and 5 others.
Measure: Number; unit: participants
Arm/Group | Benign Biliary Strictures
Number analyzed (Participants) | 23
participants
  Overall | 22
  Chronic pancreatitis (CP) | 14
  Orthotopic liver transplantation (OLT) | 3
  All others | 5

2. Primary Outcome: Long-term Success Rate in Resolution of Biliary Strictures
Description: Long-term success was defined as no clinical evidence of recurrence of the biliary stricture during the follow-up period as documented by laboratory findings or imaging and no further need for further endoscopic or surgical interventions.
Time Frame: at least 12 months after stent removal
Population: Per-protocol analysis, the 18 participants available for long term success follow-up consisted of: 11 with CP, 3 with OLT, and 4 others. Intention to treat analysis of long-term success consisted of 22 overall patients, 12 CP patients, 3 OLT patients, and 7 other patients. This analysis included all patients lost to follow-up as long-term failures.
Measure: Number; unit: participants
Groups:
- Per- Protocol Analysis of Benign Biliary Strictures: Participants underwent Endoscopic Retrograde Cholangiopancreatography (ERCP) with placement of self-expandable metal stents (SEMS) in the bile duct.
Arm/Group | Per- Protocol Analysis of Benign Biliary Strictures
Number analyzed (Participants) | 18
participants
  Overall | 15
  Chronic pancreatitis (CP) | 8
  Orthotopic liver transplantation (OLT) | 3
  All others | 4

3. Secondary Outcome: Number of Endoscopic Treatments Per Patient
Description: The average number of ERCPs performed per patient required for resolution of benign strictures.
Time Frame: At time of procedure
Measure: Mean (Full Range); unit: endoscopic treatments
Arm/Group | Benign Biliary Strictures
Number analyzed (Participants) | 23
endoscopic treatments | 2.4 [2 to 4]

4. Secondary Outcome: Ease of Stent Removal
Description: The ease of stent removal was graded on a 4-point scale (with ease, mild difficulty, significant difficulty, and failed).
Time Frame: at time of procedure
Measure: Number; unit: participants
Arm/Group | Benign Biliary Strictures
Number analyzed (Participants) | 23
participants
  With ease | 21
  Mild difficulty | 0
  Significant difficulty | 2
  Failed | 0

5. Secondary Outcome: Frequency and Severity of Adverse Events (Including Stent Migration)
Description: Adverse events were defined and graded using the 2010 American Society for Gastrointestinal Endoscopy consensus criteria
Time Frame: up to 12 months
Population: Stent migration was seen in 9/23 patients (5 downstream, 4 upstream). It was without clinical complications except in one case. Post-procedure pain experienced by 1 patient was effectively treated by downgrading the stent size to a smaller diameter.
Measure: Number; unit: participants
Arm/Group | Benign Biliary Strictures
Number analyzed (Participants) | 23
participants
  Downstream Stent Migration | 5
  Postprocedure pain due to expansion force of SEMS | 1
  Complications during stent placement | 0
  Complications during stent removal | 0
  upstream stent migration | 4

ADVERSE EVENTS:
Time Frame: 7.5 months
Description: Stent migration
Arm/Group | Benign Biliary Strictures
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 9/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benign Biliary Strictures (N=23)
stent migration (Gastrointestinal disorders) | 9 (9) — 9 subjects (39.1% of participants) had stent migration and required additional endoscopy to remove the stent
abdominal pain (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Fifty-six percent of our patients had prior therapy for their benign biliary stricture; therefore they were not treatment naive. High prevalence of CP-related strictures which are known to be more difficult to treat.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes